CLINICAL TRIAL: NCT01878617
Title: A Clinical and Molecular Risk-Directed Therapy for Newly Diagnosed Medulloblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Genentech, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJMB12; NCI-2013-01125 (Registry Identifier: NCI Clinical Trials Reporting Program); R01CA187079 (NIH)
Record Dates: First submitted 2013-06-10; First posted 2013-06-17 (Estimated); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Medulloblastoma
Keywords: SJMB12; Brain Cancer; Brain Tumors in Children; Cisplatin; Cyclophosphamide; Embryonal Tumors of CNS; GDC-0449; Gemcitabine; Hedgehog Pathway Inhibitor; Infratentorial; Mass in Brain; Medulloblastoma; Medulloblastoma Brain Tumor; Medulloblastoma Tumor; Molecular; Neuroectodermal Tumor, Primitive; Newly Diagnosed Childhood Medulloblastoma; Non-SHH Non-WNT; Pediatric Brain Tumor; Pemetrexed; Posterior Fossa Tumor; Proton Beam Therapy; Radiation Therapy; Rare Brain Tumor; Risk; SHH; Sonic Hedgehog Pathway; St Jude Medullo; St. Jude Brain Tumor Studies; St. Jude Medullo; St. Jude Studies; St. Jude Treatment; Treatment for Brain Tumors in Children; Untreated Childhood Medulloblastoma; Vincristine; Vismodegib; WNT
MeSH Terms: conditions — Medulloblastoma; Brain Neoplasms; Neuroectodermal Tumors, Primitive; Infratentorial Neoplasms | interventions — Craniospinal Irradiation; Radiotherapy; Cyclophosphamide; Cisplatin; Vincristine; HhAntag691; Pemetrexed; Gemcitabine; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Stratum W1: Low Risk (Experimental): Participants in stratum W1 will undergo reduced dose Craniospinal Irradiation with boost to the primary tumor site once daily 5 days a week for 6 weeks. Six weeks after completion of radiotherapy, patients receive one cycle of chemotherapy (cisplatin, vincristine, cyclophosphamide) once every 4 weeks for 4 cycles in absence of unacceptable toxicity. Some participants will complete aerobic training and/or neurocognitive remediation.
  Interventions: Radiation: Craniospinal Irradiation with boost to the primary tumor site; Drug: Cyclophosphamide; Drug: Cisplatin; Drug: Vincristine; Other: Aerobic Training; Other: Neurocognitive Remediation
- Stratum W2: Atypical (Experimental): Participants in stratum W2 will undergo standard dose craniospinal radiation with boost to the primary tumor site once daily 5 days a week for 6 weeks. Six weeks after completion of radiotherapy, patients receive one cycle of chemotherapy (cisplatin, vincristine, cyclophosphamide) once every 4 weeks for 4 cycles in absence of unacceptable toxicity. Some participants will complete aerobic training and/or neurocognitive remediation.
  Interventions: Radiation: Craniospinal Irradiation with boost to the primary tumor site; Drug: Cyclophosphamide; Drug: Cisplatin; Drug: Vincristine; Other: Aerobic Training; Other: Neurocognitive Remediation
- Stratum W3: High Risk (Experimental): Participants in stratum W3 will undergo high dose craniospinal radiation with boost to the primary tumor site once daily 5 days a week for 6 weeks. Six weeks after completion of radiotherapy, patients receive one cycle of chemotherapy (cisplatin, vincristine, cyclophosphamide) once every 4 weeks for 4 cycles in absence of unacceptable toxicity. Some participants will complete aerobic training and/or neurocognitive remediation.
  Interventions: Radiation: Craniospinal Irradiation with boost to the primary tumor site; Drug: Cyclophosphamide; Drug: Cisplatin; Drug: Vincristine; Other: Aerobic Training; Other: Neurocognitive Remediation
- Stratum S1: Standard Risk (Experimental): Participants in stratum S1 will undergo standard dose craniospinal radiation with boost to the primary tumor site once daily 5 days a week for 6 weeks. Six weeks after completion of radiotherapy, patients receive one cycle of chemotherapy (cisplatin, vincristine, cyclophosphamide) once every 4 weeks for 4 cycles in absence of unacceptable toxicity. After completion of 4 cycles of chemotherapy, participants who are skeletally mature will receive maintenance chemotherapy with vismodegib. Some participants will complete aerobic training and/or neurocognitive remediation.
  Interventions: Radiation: Craniospinal Irradiation with boost to the primary tumor site; Drug: Cyclophosphamide; Drug: Cisplatin; Drug: Vincristine; Drug: Vismodegib; Other: Aerobic Training; Other: Neurocognitive Remediation
- Stratum S2: High Risk (Experimental): Participants in stratum S2 will undergo high dose craniospinal radiation with boost to the primary tumor site once daily 5 days a week for 6 weeks. Six weeks after completion of radiotherapy, patients receive one cycle of chemotherapy (cisplatin, vincristine, cyclophosphamide) once every 4 weeks for 4 cycles in absence of unacceptable toxicity. After completion of 4 cycles of chemotherapy, participants who are skeletally mature will receive maintenance chemotherapy with vismodegib. Some participants will complete aerobic training and/or neurocognitive remediation.
  Interventions: Radiation: Craniospinal Irradiation with boost to the primary tumor site; Drug: Cyclophosphamide; Drug: Cisplatin; Drug: Vincristine; Drug: Vismodegib; Other: Aerobic Training; Other: Neurocognitive Remediation
- Stratum N1: Standard Risk (Experimental): Participants in stratum N1 will undergo standard dose craniospinal radiation with boost to the primary tumor site once daily 5 days a week for 6 weeks. Six weeks after completion of radiotherapy, patients receive one cycle of chemotherapy (cisplatin, vincristine, cyclophosphamide) once every 4 weeks for 4 cycles in absence of unacceptable toxicity. Some participants will complete aerobic training and/or neurocognitive remediation.
  Interventions: Radiation: Craniospinal Irradiation with boost to the primary tumor site; Drug: Cyclophosphamide; Drug: Cisplatin; Drug: Vincristine; Other: Aerobic Training; Other: Neurocognitive Remediation
- Stratum N2: Intermediate Risk (Experimental): Participants in stratum N2 will undergo standard dose craniospinal radiation with boost to the primary tumor site once daily 5 days a week for 6 weeks. Six weeks after completion of radiotherapy, patients receive standard chemotherapy (cisplatin, vincristine, cyclophosphamide) for 4 cycles intermixed with an additional 3 cycles of chemotherapy with pemetrexed and gemcitabine in absence of unacceptable toxicity. Some participants will complete aerobic training and/or neurocognitive remediation.
  Interventions: Radiation: Craniospinal Irradiation with boost to the primary tumor site; Drug: Cyclophosphamide; Drug: Cisplatin; Drug: Vincristine; Drug: Pemetrexed; Drug: Gemcitabine; Other: Aerobic Training; Other: Neurocognitive Remediation
- Stratum N3: High Risk (Experimental): Participants in stratum N3 will undergo high dose craniospinal radiation with boost to the primary tumor site once daily 5 days a week for 6 weeks. Six weeks after completion of radiotherapy, patients receive standard chemotherapy (cisplatin, vincristine, cyclophosphamide) for 4 cycles intermixed with an additional 3 cycles of chemotherapy with pemetrexed and gemcitabine in absence of unacceptable toxicity. Some participants will complete aerobic training and/or neurocognitive remediation.
  Interventions: Radiation: Craniospinal Irradiation with boost to the primary tumor site; Drug: Cyclophosphamide; Drug: Cisplatin; Drug: Vincristine; Drug: Pemetrexed; Drug: Gemcitabine; Other: Aerobic Training; Other: Neurocognitive Remediation

INTERVENTIONS:
Radiation: Craniospinal Irradiation with boost to the primary tumor site — All participants will undergo craniospinal irradiation (CSI) with boost to the primary tumor site. The dose given is based on the molecular and risk group as noted in the arm descriptions. The type of radiation used includes conformal radiation therapy (photons) or intensity modulated radiation therapy (IMRT) or proton beam therapy.
  Other Names: CSI; Radiation treatments
Drug: Cyclophosphamide — Route of Administration (ROA): Intravenously (IV)
  Other Names: Cytoxan(R)
Drug: Cisplatin — ROA: IV
  Other Names: Platinol-AQ(R)
Drug: Vincristine — ROA: IV
  Other Names: Oncovin(R)
Drug: Vismodegib — ROA: Orally (PO)
  Other Names: Erivedge(TM); GDC-0449
  Arms: Stratum S1: Standard Risk; Stratum S2: High Risk
Drug: Pemetrexed — ROA: IV
  Other Names: Almita(R)
  Arms: Stratum N2: Intermediate Risk; Stratum N3: High Risk
Drug: Gemcitabine — ROA: IV
  Other Names: Gemzar
  Arms: Stratum N2: Intermediate Risk; Stratum N3: High Risk
Other: Aerobic Training
  Other Names: Exercise
Other: Neurocognitive Remediation
  Other Names: Computer-based working memory intervention; Cogmed

SUMMARY:
Historically, medulloblastoma treatment has been determined by the amount of leftover disease present after surgery, also known as clinical risk (standard vs. high risk). Recent studies have shown that medulloblastoma is made up of distinct molecular subgroups which respond differently to treatment. This suggests that clinical risk alone is not adequate to identify actual risk of recurrence. In order to address this, we will stratify medulloblastoma treatment in this phase II clinical trial based on both clinical risk (low, standard, intermediate, or high risk) and molecular subtype (WNT, SHH, or Non-WNT Non-SHH). This stratified clinical and molecular treatment approach will be used to evaluate the following:

* To find out if participants with low-risk WNT tumors can be treated with a lower dose of radiation to the brain and spine, and a lower dose of the chemotherapy drug cyclophosphamide while still achieving the same survival rate as past St. Jude studies with fewer side effects.
* To find out if adding targeted chemotherapy after standard chemotherapy will benefit participants with SHH positive tumors.
* To find out if adding new chemotherapy agents to the standard chemotherapy will improve the outcome for intermediate and high risk Non-WNT Non-SHH tumors.
* To define the cure rate for standard risk Non-WNT Non-SHH tumors treated with reduced dose cyclophosphamide and compare this to participants from the past St. Jude study.

All participants on this study will have surgery to remove as much of the primary tumor as safely possible, radiation therapy, and chemotherapy. The amount of radiation therapy and type of chemotherapy received will be determined by the participant's treatment stratum. Treatment stratum assignment will be based on the tumor's molecular subgroup assignment and clinical risk.

The participant will be assigned to one of three medulloblastoma subgroups determined by analysis of the tumor tissue for tumor biomarkers:

* WNT (Strata W): positive for WNT biomarkers
* SHH (Strata S): positive for SHH biomarkers
* Non-WNT Non-SHH, Failed, or Indeterminate (Strata N): negative for WNT and SHH biomarkers or results are indeterminable

Participants will then be assigned to a clinical risk group (low, standard, intermediate, or high) based on assessment of:

* How much tumor is left after surgery
* If the cancer has spread to other sites outside the brain [i.e., to the spinal cord or within the fluid surrounding the spinal cord, called cerebrospinal fluid (CSF)]
* The appearance of the tumor cells under the microscope
* Whether or not there are chromosomal abnormalities in the tumor, and if present, what type (also called cytogenetics analysis)

DETAILED DESCRIPTION:
Primary Objectives:

* To estimate the progression free survival distribution of WNT-medulloblastoma patients treated on Stratum W1 with reduced-dose craniospinal irradiation and reduced-dose cyclophosphamide.
* To estimate progression-free survival distribution of Non-WNT Non-SHH medulloblastoma patients treated on Stratum N1 with reduced dose cyclophosphamide.
* To estimate the progression free survival distribution of skeletally mature SHH medulloblastoma patients assigned to Stratum S1 and treated with oral maintenance therapy using a targeted SHH pathway inhibitor (vismodegib) after the adjuvant chemotherapy regimen is complete and to compare the outcome to molecularly and clinically matched historical controls from SJMB03 as well as outcome from other published cohorts.
* To evaluate the effect of an aerobic training intervention, delivered during the radiation therapy period and at home, prior to the start of chemotherapy, on cardiopulmonary fitness.
* To assess the impact of a computer-based working memory intervention (administered prophylactically at the end of chemotherapy), relative to standard of care, on a performance-based measure of working memory.

Secondary Objectives:

* To estimate overall survival distribution of WNT-medulloblastoma patients treated on Stratum W1 with reduced-dose craniospinal irradiation and reduced-dose cyclophosphamide and compare progression free and overall survival distributions to molecularly and clinically matched historical controls from St. Jude SJMB03 study.
* To estimate the progression free (in S1 skeletally immature and S2 both sub-strata) and overall survival distributions of SHH medulloblastoma patients enrolled on Strata S1 and S2 some of whom will be treated with oral maintenance therapy using a targeted SHH pathway inhibitor (vismodegib) after adjuvant chemotherapy regimen is complete and compare these outcomes to molecularly and clinically matched historical controls from SJMB03 as well as outcome from other published cohorts.
* To estimate the progression free and overall survival distributions of Non-WNT Non-SHH medulloblastoma patients treated on Strata N2 and N3 with 3 cycles of pemetrexed and gemcitabine in addition to 4 cycles of conventional adjuvant chemotherapy and compare the progression-free and overall survival distributions to molecularly and clinically matched historical controls from St. Jude SJMB03 study separately for each stratum.
* To estimate the overall survival distribution of Non-WNT Non-SHH medulloblastoma patients treated on Stratum N1 with reduced dose cyclophosphamide and compare progression free and overall survival distributions to molecularly and clinically matched historical controls from St. Jude SJMB03 study.
* To evaluate the feasibility and toxicity of adding pemetrexed and gemcitabine to adjuvant chemotherapy regimen of intermediate and high risk Non-WNT Non-SHH medulloblastoma patients (Strata N2 and N3).
* To evaluate the feasibility and toxicity of oral maintenance therapy with the targeted SHH inhibitor (vismodegib) after conventional adjuvant chemotherapy regimen is complete.
* To estimate the cumulative incidence of local disease failure at 2 and 5 years based on treatment regimen, strata, and clinical and treatment factors.
* To evaluate the effects of an aerobic training intervention, delivered during the radiation therapy period and at home, prior to the start of chemotherapy, on physical performance, fatigue, health related quality of life, memory, attention and executive function at the end of the intervention, at the end of adjuvant chemotherapy, and one, two and five years off adjuvant chemotherapy, among children treated for medulloblastoma.
* To evaluate the impact of an aerobic training intervention on sleep quality and quantity in children with medulloblastoma.
* To evaluate the relation between baseline cognitive performance and the variables of sleep quality and quantity, and fatigue in children with medulloblastoma.
* To estimate change in neurocognitive performance using a comprehensive assessment battery (e.g., measures of intellectual function, academic abilities, attention, memory, processing speed and executive functions) and investigate the relationship of change to relevant demographic factors (e.g., gender, age at treatment, time since treatment and socioeconomic status) and clinical factors (e.g., treatment intensity/risk group, posterior fossa syndrome).
* To assess the impact of a computer-based working memory intervention, relative to standard of care, on additional performance- and rater-based measures of attention, processing speed and executive functions.
* To compare the impact of a computer-based working memory intervention in conjunction with an aerobic training intervention, relative to either intervention in isolation, on measures of attention, processing speed and executive functions.
* To evaluate the maintenance of improvements on measures of attention, working memory, processing speed and executive functions six months following participation in the computer-based working memory intervention program.

Outline: This is a multicenter study. Patients are stratified according to molecular subgroup assignment (WNT, SHH, or Non-WNT Non- SHH) and then by clinical risk stratification (extent of resection, M stage, histologic subtype, and cytogenetic features). All patients will be treated with risk-adapted radiation therapy and adjuvant chemotherapy. Patients assigned to Stratum W1 will receive reduced dose radiation therapy. Patients assigned to Stratum W2, S1, N1, or N2 will receive standard dose radiation therapy. Patients assigned to Stratum W3, S2, or N3 will receive high dose radiation therapy. Radiation therapy will be followed by 4 cycles of adjuvant conventional chemotherapy with cyclophosphamide, cisplatin and vincristine for all patients. Patients assigned to Stratum N2 or N3 (Non-WNT Non-SHH with high risk factors) will receive 3 additional cycles of pemetrexed and gemcitabine chemotherapy intermixed into the conventional adjuvant chemotherapy cycles. Patients with SHH subtype (Stratum S1 or S2) who are skeletally mature will receive 12 months additional maintenance therapy with vismodegib.

Patients may consent to provide tumor tissue, blood, and CSF samples for biological studies. Tumor tissues are analyzed for the activation of the WNT signaling pathway, activation of the SHH signaling pathway, validation of novel patterns of gene expression via immunohistochemical (IHC) analysis; validation of genetic abnormalities via interphase fluorescence in situ hybridization (iFISH); construction of gene expression profiles via microarray analysis; construction of DNA methylation profiling via microarrays; single nucleotide polymorphism (SNP) analysis for DNA copy number aberrations; potential oncogenes and tumor suppressor genes via DNA sequence analysis; expression of a number of cell signal proteins implicated in the biology of medulloblastoma via western blot; expression of additional proteins encoded by genes associated through SNP and gene expression array analysis with clinical disease behavior. Blood samples are analyzed from patients whose tumors contain gene mutations via sequence analysis of constitutional DNA. CSF and blood samples are analyzed for identification of potential tumor markers. Parents may consent to have blood samples analyzed for inheritable gene mutations associated with medulloblastoma.

Patients may also consent to exploratory research that include additional functional MRI imaging to investigate damage to neural connections from therapy; additional psychological testing to identify neurocognitive effects of therapy; additional heart and lung testing to identify treatment effects; additional endocrine studies to identify treatment effect on growth and development.

After completion of study treatment, patients are followed every 6 months for 5 years.

ELIGIBILITY:
INCLUSION CRITERIA

* Medulloblastoma or medulloblastoma variants including posterior fossa PNET as documented by an institutional pathologist.
* Participant's age meets one of the following: (1) Age greater than or equal to 3 years and less than 22 years of age at the time of diagnosis (may enroll on Strata W, S or N), OR (2) age is greater than or equal to 22 years and less than 40 years AND patient has SHH medulloblastoma (must enroll on Stratum S).
* No previous radiotherapy, chemotherapy or other brain tumor directed therapy other than corticosteroid therapy and surgery.
* Patients must begin treatment as outlined in the protocol within 36 days of definitive surgery (day of surgery is day 0; definitive surgery includes second surgeries to resect residual tumor).
* Adequate performance status: children < 10-Lansky Score ≥ 30; children ≥ 10-Karnofsky ≥ 30 (except for posterior fossa syndrome).
* Females of child-bearing potential cannot be pregnant or breast-feeding. Female participants > 10 years of age or post-menarche must have a negative serum or urine pregnancy test prior to enrollment.
* Biological parent(s) of participant (child) enrolling on this protocol. These parents will be assigned to cohort P. The exclusion criteria below do not apply to this cohort.

EXCLUSION CRITERIA

* CNS embryonal tumor other than medulloblastoma or PNET in the posterior fossa, for example, patients with diagnosis of Atypical Teratoid / Rhabdoid Tumor (ATRT), supratentorial PNET, pineoblastoma, ependymoblastoma, ETANTR are excluded.
* Research participants with other clinically significant medical disorders that could compromise their ability to tolerate protocol therapy or would interfere with the study procedures or results history.

Participants in the Stratum S maintenance chemotherapy portion of the study must meet the criteria below prior to start of vismodegib therapy:

* Participants must be Stratum S (SHH)
* Participants must be skeletally mature defined as females with a bone age ≥ 15 years and males with a bone age ≥ 17 years.
* Must be able to swallow pills
* BSA must be >0.67 and <2.5 m2
* Male and female participants of reproductive potential must agree to effective contraception during and after study treatment. See Appendices I and II for further guidance for participants receiving vismodegib
* ANC ≥ 1000/mm^3 (after G-CSF discontinued)
* Platelets ≥ 50,000/mm^3 (without support)
* Hgb ≥ 8 g/dL (with or without transfusion support)
* Serum creatinine ≤ 1.5 mg/dL
* Total bilirubin ≤ 1.5X the institutional ULN
* SGPT (ALT) ≤ 2.5X the institutional ULN
* SGOT (AST) ≤ 2.5X the institutional ULN
* Alkaline Phosphatase ≤ 1.5X the institutional ULN
* Serum albumin ≥ 2.5 g/dL

Participants in the exercise intervention portion of the study must meet all criteria below:

* Must be ≥ 5 years and < 22 years at the time of enrollment
* Must have no congenital heart disease
* Must be capable of performing the exercise intervention at the time of baseline assessment as determined by the treating physician.

Participants in the cognitive remediation intervention portion of the study must meet all criteria below:

* Completed protocol-directed radiation therapy
* ≥5 years at the time of remediation intervention consent or age is greater than or equal to 22 years and less than 40 years and patient has SHH medulloblastoma
* English as primary language and training aide who speaks English available to participate in required sessions
* No significant cognitive impairment operationalized as either an IQ < 70 for children with St. Jude SJMB12 study baseline testing or based on clinician judgment baseline IQ missing
* No major sensory or motor impairment that would preclude valid cognitive testing (e.g., unresolved posterior fossa syndrome, blindness, poorly controlled seizures/photosensitive epilepsy, psychosis) or a major psychological condition that would preclude completion of the intervention (e.g., significant oppositionality, autism spectrum disorder, severe anxiety or depressive symptoms)

Ages: 3 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 660 (Actual)
Dates: Start 2013-06-23 (Actual); Primary Completion 2028-10-13 (Estimated); Study Completion 2031-10-13 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival in Stratum W1 | 2 years after diagnosis
  Progression-free survival (PFS) will be measured from diagnosis to the earliest of disease progression or death from any cause. Patients who have not experienced one of these events will be censored at their last date of contact.
Progression-free Survival in Stratum N1 | 2 years after diagnosis
  Progression-free survival (PFS) will be measured from diagnosis to the earliest of disease progression or death from any cause. Patients who have not experienced one of these events will be censored at their last date of contact.
Progression-free Survival in Stratum S1 Skeletally Mature Cohort | 2 years after diagnosis
  Progression-free survival (PFS) will be measured from diagnosis to the earliest of disease progression or death from any cause. Patients who have not experienced one of these events will be censored at their last date of contact. PFS in SJMB12 stratum S1 skeletally mature cohort will be compared to historical controls from SJMB03 as well as from another published cohort (Thompson et al., 2016) using log-rank test.
Change in VO2 Peak Value | baseline and 12 weeks post-randomization
  To evaluate the effect of an aerobic training intervention on cardiopulmonary fitness.
Change in Spatial Span Backward Standard Score | baseline and 10-12 weeks post baseline
  To assess the impact of a computer-based working memory intervention, relative to standard of care, on a performance-based measure of working memory.

SECONDARY OUTCOMES:
Progression-free Survival in Stratum W1 Compared to Historical Controls | 2 years after diagnosis
  Progression-free survival (PFS) in stratum W1 will be compared to historical controls from SJMB03 using log-rank test.
Overall Survival in Stratum W1 | 2 years after diagnosis
  Overall survival (OS) will be measured from diagnosis to death from any cause. Patients who survive will be censored at their last date of contact. OS in SJMB12 stratum W1 will be compared to historical controls from SJMB03 using log-rank test.
Progression-free Survival in Stratum S1 Skeletally Immature Cohort | 2 years after diagnosis
  Progression-free survival (PFS) will be measured from diagnosis to the earliest of disease progression or death from any cause. Patients who have not experienced one of these events will be censored at their last date of contact. PFS in SJMB12 stratum S1 skeletally immature cohort will be compared to historical controls from SJMB03 as well as from another published cohort (Thompson et al., 2016) using log-rank test.
Progression-free Survival in Stratum S2 Skeletally Mature Cohort | 2 years after diagnosis
  Progression-free survival (PFS) will be measured from diagnosis to the earliest of disease progression or death from any cause. Patients who have not experienced one of these events will be censored at their last date of contact. PFS in SJMB12 stratum S2 skeletally mature cohort will be compared to historical controls from SJMB03 as well as from another published cohort (Thompson et al., 2016) using log-rank test.
Progression-free Survival in Stratum S2 Skeletally Immature Cohort | 2 years after diagnosis
  Progression-free survival (PFS) will be measured from diagnosis to the earliest of disease progression or death from any cause. Patients who have not experienced one of these events will be censored at their last date of contact. PFS in SJMB12 stratum S2 skeletally immature cohort will be compared to historical controls from SJMB03 as well as from another published cohort (Thompson et al., 2016) using log-rank test.
Overall Survival in Stratum S1 Skeletally Mature Cohort | 2 years after diagnosis
  Overall survival (OS) will be measured from diagnosis to death from any cause. Patients who survive will be censored at their last date of contact. OS in SJMB12 stratum S1 skeletally mature cohort will be compared to historical controls from SJMB03 as well as from another published cohort (Thompson et al., 2016) using log-rank test.
Overall Survival in Stratum S1 Skeletally Immature Cohort | 2 years after diagnosis
  Overall survival (OS) will be measured from diagnosis to death from any cause. Patients who survive will be censored at their last date of contact. OS in SJMB12 stratum S1 skeletally immature cohort will be compared to historical controls from SJMB03 as well as from another published cohort (Thompson et al., 2016) using log-rank test.
Overall Survival in Stratum S2 Skeletally Mature Cohort | 2 years after diagnosis
  Overall survival (OS) will be measured from diagnosis to death from any cause. Patients who survive will be censored at their last date of contact. OS in SJMB12 stratum S2 skeletally mature cohort will be compared to historical controls from SJMB03 as well as from another published cohort (Thompson et al., 2016) using log-rank test.
Overall Survival in Stratum S2 Skeletally Immature Cohort | 2 years after diagnosis
  Overall survival (OS) will be measured from diagnosis to death from any cause. Patients who survive will be censored at their last date of contact. OS in SJMB12 stratum S2 skeletally immature cohort will be compared to historical controls from SJMB03 as well as from another published cohort (Thompson et al., 2016) using log-rank test.
Progression-free Survival in Stratum N2 | 2 years after diagnosis
  Progression-free survival (PFS) will be measured from diagnosis to the earliest of disease progression or death from any cause. Patients who have not experienced one of these events will be censored at their last date of contact. PFS in SJMB12 stratum N2 will be compared to historical controls from SJMB03 using log-rank test.
Overall Survival in Stratum N2 | 2 years after diagnosis
  Overall survival (OS) will be measured from diagnosis to death from any cause. Patients who survive will be censored at their last date of contact. OS in SJMB12 stratum N2 will be compared to historical controls from SJMB03 using log-rank test.
Progression-free Survival in Stratum N3 | 2 years after diagnosis
  Progression-free survival (PFS) will be measured from diagnosis to the earliest of disease progression or death from any cause. Patients who have not experienced one of these events will be censored at their last date of contact. PFS in SJMB12 stratum N3 will be compared to historical controls from SJMB03 using log-rank test.
Overall Survival in Stratum N3 | 2 years after diagnosis
  Overall survival (OS) will be measured from diagnosis to death from any cause. Patients who survive will be censored at their last date of contact. OS in SJMB12 stratum N3 will be compared to historical controls from SJMB03 using log-rank test.
Progression-free Survival in Stratum N1 Compared to Historical Controls | 2 years after diagnosis
  Progression-free survival (PFS) in stratum N1 will be compared to historical controls from SJMB03 using log-rank test.
Overall Survival in Stratum N1 | 2 years after diagnosis
  Overall survival (OS) will be measured from diagnosis to death from any cause. Patients who survive will be censored at their last date of contact. OS in SJMB12 stratum N1 will be compared to historical controls from SJMB03 using log-rank test.
Percentage of Participants Who Complete Pemetrexed and Gemcitabine Therapy | 10 months after on treatment
  Intermediate and high risk Non-WNT Non-SHH medulloblastoma patients treated on strata N2 and N3 will receive pemetrexed and gemcitabine during adjuvant chemotherapy. Percentage of participants who complete treatment will be estimated and reported with an exact 2-sided 95% confidence interval.
Percentage of Participants Who Complete Vismodegib Therapy | 20 months after on treatment
  Patients with SHH tumor treated on strata S1 and S2 will receive 12 courses of vismodegib during maintenance therapy. For each risk-based stratum separately, percentage of participants who complete treatment will be estimated and reported with an exact 2-sided 95% confidence interval.
Number of Local Failures | 2 and 5 years after on treatment
  To estimate stratum specific cumulative incidence of local disease failure at 2 and 5 years.
Change in hand grip strength | Baseline (at enrollment), 12 weeks, at end of adjuvant chemotherapy (28 weeks for strata W1/W2/W3/N1/S1/S2 and 40 weeks for strata N2/N3), and 1, 2, and 5 years after the last patient enrollment
  To evaluate the effects of an aerobic training intervention, delivered during the radiation therapy period and at home, prior to the start of chemotherapy, on hand grip strength as measured using a hand-held dynamometer among children treated for medulloblastoma. Participants will be seated with the shoulder at 0-10 degrees and the elbow in 90 degrees of flexion. The forearm will be positioned in neutral. Each participant will complete three trials, the average used for analysis.
Change in range of motion | Baseline (at enrollment), 12 weeks, at end of adjuvant chemotherapy (28 weeks for strata W1/W2/W3/N1/S1/S2 and 40 weeks for strata N2/N3), and 1, 2, and 5 years after the last patient enrollment
  To evaluate the effects of an aerobic training intervention, delivered during the radiation therapy period and at home, prior to the start of chemotherapy, on range of motion as measured with a goniometer among children treated for medulloblastoma. The goniometer is a reliable and valid measure of active and passive range of motion with standard procedures.
Change in overall flexibility | Baseline (at enrollment), 12 weeks, at end of adjuvant chemotherapy (28 weeks for strata W1/W2/W3/N1/S1/S2 and 40 weeks for strata N2/N3), and 1, 2, and 5 years after the last patient enrollment
  To evaluate the effects of an aerobic training intervention, delivered during the radiation therapy period and at home, prior to the start of chemotherapy, on overall flexibility among children treated for medulloblastoma. Flexibility will be measured by having participants perform a "sit and reach test." A yardstick is placed on a firm flat surface and tape is placed across it at a right angle to the 15 inch mark. The participant sits with the yardstick between the legs, with legs extended at right angles to the taped line on the floor. The heels of the feet touch the edge of the taped line and are 10-12 inches apart. The participant reaches forward with both hands as far as possible, and the best value for three trials, in centimeters, at the fingertips is recorded.
Change in motor proficiency | Baseline (at enrollment), 12 weeks, at end of adjuvant chemotherapy (28 weeks for strata W1/W2/W3/N1/S1/S2 and 40 weeks for strata N2/N3), and 1, 2, and 5 years after the last patient enrollment
  Measured by the Bruininks-Oseretsky Test of Motor Proficiency, Version 2 (BOT-2). To evaluate the effects of an aerobic training intervention, delivered during the radiation therapy period and at home, prior to the start of chemotherapy, on motor proficiency among children treated for medulloblastoma.
Change in quality of life (QOL) score | Baseline (at enrollment), 12 weeks, at end of adjuvant chemotherapy (28 weeks for strata W1/W2/W3/N1/S1/S2 and 40 weeks for strata N2/N3), and 1, 2, and 5 years after the last patient enrollment
  To evaluate the effects of an aerobic training intervention, delivered during the radiation therapy period and at home, prior to the start of chemotherapy on health related quality of life (QoL) among children treated for medulloblastoma. QoL will be assessed using the 23-item PedsQL(TM) 4.0 Generic Core Scales which encompasses four subscales (1) physical functioning (eight items), (2) emotional functioning (five items), (3) social functioning (five items), and (4) school functioning (five items) and the 24-item PedsQL(TM) Brain Tumor Module which encompasses six scales: (1) cognitive problems (seven items), (2) pain and hurt (three items), (3) movement and balance (three items), (4) procedural anxiety (three items), (5) nausea (five items), and (6) worry (three items).
Change in fatigue score | Baseline (at enrollment), 12 weeks, at end of adjuvant chemotherapy (28 weeks for strata W1/W2/W3/N1/S1/S2 and 40 weeks for strata N2/N3), and 1, 2, and 5 years after the last patient enrollment
  To evaluate the effects of an aerobic training intervention, delivered during the radiation therapy period and at home, prior to the start of chemotherapy, on fatigue among children treated for medulloblastoma. Fatigue will be assessed using the 18-item PedsQL(TM) Multidimensional Fatigue Scale which encompasses three subscales: (1) general fatigue (six items), (2) sleep/rest fatigue (six items), and (3) cognitive fatigue (six items).
Change in measure of memory function | Baseline (at enrollment), 12 weeks, and at end of adjuvant chemotherapy (28 weeks for strata W1/W2/W3/N1/S1/S2 and 40 weeks for strata N2/N3).
  To evaluate the effects of an aerobic training intervention, delivered during the radiation therapy period and at home, prior to the start of chemotherapy, on memory function at the end of the intervention and at the end of adjuvant chemotherapy, among children treated for medulloblastoma. Memory will be measured using different instruments as age appropriate: CogStage for age 5 and older (Continuous Paired Associate Learning task), California Verbal Learning Test, Children's Version (CVLT-C) for age 6 to < 17 years or California Verbal Learning Test, Second Edition (CVLT-II) for age ≥17 years.
Change in measure of attention | Baseline (at enrollment), 12 weeks, and at end of adjuvant chemotherapy (28 weeks for strata W1/W2/W3/N1/S1/S2 and 40 weeks for strata N2/N3).
  To evaluate the effects of an aerobic training intervention, delivered during the radiation therapy period and at home, prior to the start of chemotherapy, on attention at the end of the intervention and at the end of adjuvant chemotherapy, among children treated for medulloblastoma. Attention will be measured using different instruments as age appropriate: Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) for ages 3 to < 6 years (Digit Span Forward subtest), Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV) for ages 6 to < 17 years (Digit Span Forward subtest) or Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) for ages ≥17 years (Digit Span Forward subtest). We will also use Conners' Continuous Performance Test, Kiddie Version V.5 for ages 4 to < 6 years and Conner's Continuous Performance Test, Second Edition (CPT-II) for ages ≥6 years, in addition to Cog Stage for children ≥5 years (Detection and Identification tasks).
Change in executive function score | Baseline (at enrollment), 12 weeks, and at end of adjuvant chemotherapy (28 weeks for strata W1/W2/W3/N1/S1/S2 and 40 weeks for strata N2/N3).
  To evaluate the effects of an aerobic training intervention, delivered during the radiation therapy period and at home, prior to the start of chemotherapy, on executive function at the end of the intervention and at the end of adjuvant chemotherapy, among children treated for medulloblastoma. Executive function is measured as age-appropriate by the following: BRIEF-P (age 3 to <6 years), BRIEF (age 6 to <19 years) and BREIF-A (age ≥19 years). Connor's Parent Rating Scale, Third Edition (CPRS-III) will also be used for age 6 to <19 years, as well as CogState One-Back and Groton Maze tasks for age ≥5 years.
Change in sleep | Baseline and 10-12 weeks post randomization
  To evaluate the impact of an aerobic training intervention on sleep quality and quantity in children with medulloblastoma. Sleep quality and quantity will be measured by Actigraph accelerometer as well as a sleep diary.
Association between baseline cognitive performance and sleep quality | Baseline and approximately 7-10 months after treatment
  To evaluate the relation between baseline cognitive performance and sleep quality in children with medulloblastoma. Multivariable general linear mixed models will be used to look for associations between sleep quality as measured by Actigraph accelerometer and a sleep diary with measures of cognitive performance (memory, attention and executive function (detailed above) and internalizing and externalizing behavior. Internalizing and externalizing behaviors will be measured using the Behavior Assessment System for Children, 2nd Edition (BASC-2). There are Preschool, Child and Adolescent versions.
Association between baseline cognitive performance and sleep quantity | Baseline and approximately 7-10 months after treatment
  To evaluate the relation between baseline cognitive performance and sleep quantity in children with medulloblastoma. Multivariable general linear mixed models will be used to look for associations between sleep quantity as measured by a sleep diary with measures of cognitive performance (memory, attention and executive function and internalizing and externalizing behavior (detailed above).
Association between baseline cognitive performance and fatigue | Baseline and approximately 7-10 months after treatment
  To evaluate the relation between baseline cognitive performance and fatigue in children with medulloblastoma. Multivariable general linear mixed models will be used to look for associations between fatigue score as measured by the Multidimensional Fatigue Scale with measures of cognitive performance (memory, attention and executive function and internalizing and externalizing behavior (detailed above).
Longitudinal change in measure of intellectual function | Baseline through 5 years after enrollment
  Intellectual function will be measured as age-appropriate using the Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) for age 3 to < 6 years, Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV) for age 6 to < 17 years, and Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) for age ≥17 years. Linear mixed-effects models will be used to model change in intellectual function over time.
Association of demographic and clinical factors with change in intellectual function | Baseline through 5 years after enrollment
  Intellectual function will be measured as age-appropriate using the Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) for age 3 to < 6 years, Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV) for age 6 to < 17 years, and Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) for age ≥17 years. Linear mixed-effects models and multivariate linear mixed-effects models will be used to examine change in intellectual function with demographic and clinical factors.
Longitudinal change in measure of academic ability | Baseline through 5 years after enrollment
  Academic ability will be measured using the Woodcock Johnson Tests of Academic Achievement-Third Edition (WJ-III-ACH) which has six subsets: Letter-Word Identification, Passage Comprehension, Reading Fluency, Calculation, Applied Problems, and Math Fluency. Academic ability will also be measured using the Comprehensive Test of Phonological Processing (CTOPP) which has three subsets: Elision, Blending Words, and Rapid Naming. Linear mixed-effects models will be used to model change in academic ability over time.
Association of demographic and clinical factors with change in academic ability | Baseline through 5 years after enrollment
  Linear mixed-effects models and multivariate linear mixed-effects models will be used to examine change in academic ability (measured as described above) with demographic and clinical factors.
Longitudinal change in measure of attention | Baseline through 5 years after enrollment
  Attention will be measured using different instruments as age appropriate: Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) for ages 3 to < 6 years old (Digit Span Forward subtest), Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV) for ages 6 to < 17 years (Digit Span Forward subtest) or Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) for ages ≥17 years (Digit Span Forward subtest). We will also use Conners' Continuous Performance Test, Kiddie Version V.5 for ages 4 to < 6 years and Conner's Continuous Performance Test, Second Edition (CPT-II) for ages ≥6 years, in addition to Cog Stage for children ≥5 years (Detection and Identification tasks). Linear mixed-effects models will be used to model change in the measure of attention over time.
Association of demographic and clinical factors with change in attention | Baseline through 5 years after enrollment
  Linear mixed-effects models and multivariate linear mixed-effects models will be used to examine change in attention (measured as described above) with demographic and clinical factors.
Longitudinal change in measure of memory | Baseline through 5 years after enrollment
  Memory will be measured using different instruments as age appropriate: CogStage for age 5 and older (Continuous Paired Associate Learning task), California Verbal Learning Test, Children's Version (CVLT-C) for age 6 to < 17 years or California Verbal Learning Test, Second Edition (CVLT-II) for age ≥17 years. Linear mixed-effects models will be used to model change in memory over time.
Association of demographic and clinical factors with change in memory | Baseline through 5 years after enrollment
  Linear mixed-effects models and multivariate linear mixed-effects models will be used to examine change in memory (measured as described above) with demographic and clinical factors.
Longitudinal change in measure of cognitive processing speed function | Baseline through 5 years after enrollment
  Cognitive processing speed function will be measured using the age-appropriate processing speed indices: WPPSI-IV which has two subsets: Bug Search and Cancellation, for age 3 to < 6 years old; WISC-IV which has two subsets: Coding and Symbol Search subtests, for 6 to < 17 years, and WAIS-IV which has two subsets: Coding and Symbol Search subtests, for age ≥17 years. Linear mixed-effects models will be used to model change in cognitive processing speed over time.
Association of demographic and clinical factors with change in cognitive processing speed | Baseline through 5 years after enrollment
  Linear mixed-effects models and multivariate linear mixed-effects models will be used to examine change in cognitive processing speed (measured as described above) with demographic and clinical factors.
Longitudinal change in measure of neurocognitive executive function | Baseline through 5 years after enrollment
  Neurocognitive executive function will be measured using the Behavioral rating inventory of executive function (BRIEF). There are age-appropriate versions: BRIEF-P for age 3 to < 6 years, BRIEF for age 6 to <19 years, and BRIEF-A for age ≥19 years. Executive function will also be measured using Conner's Parent Rating Scale, Third Edition (CPRS-III), for age 6 to < 19 years and also CogState, for age ≥5 years, One-Back and Groton Maze tasks. Linear mixed-effects models will be used to model change in executive function over time.
Association of demographic and clinical factors with change in neurocognitive executive function | Baseline through 5 years after enrollment
  Linear mixed-effects models and multivariate linear mixed-effects models will be used to examine change in executive function (measured as described above) with demographic and clinical factors.
Change in measure of attention | Baseline (at 7-10 months after start of therapy) and at 3 months after baseline
  To assess the impact of a computer-based working memory intervention, relative to standard of care, on additional performance- and rater-based measure of attention. Attention will be measured using different instruments as age appropriate: Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) for ages 3 to < 6 years (Digit Span Forward subtest), Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV) for ages 6 to < 17 years (Digit Span Forward subtest) or Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) for ages ≥17 years (Digit Span Forward subtest). We will also use Conners' Continuous Performance Test, Kiddie Version V.5 for ages 4 to < 6 years and Conner's Continuous Performance Test, Second Edition (CPT-II) for ages ≥6 years, in addition to Cog Stage for children ≥5 years (Detection and Identification tasks). T tests will be used to compare changes in attention between the intervention and standard of care groups.
Change in measure of processing speed | Baseline (at 7-10 months after start of therapy) and at 3 months after baseline
  To assess the impact of a computer-based working memory intervention, relative to standard of care, on additional performance- and rater-based measure of processing speed. Cognitive processing speed function will be measured using the age-appropriate processing speed indices: WPPSI-IV which has two subsets: Bug Search and Cancellation, for age 3 to < 6 years; WISC-IV which has two subsets: Coding and Symbol Search subtests, for 6 to < 17 years, and WAIS-IV which has two subsets: Coding and Symbol Search subtests, for age ≥17 years. T tests will be used to compare changes in processing speed between the intervention and standard of care groups.
Change in measure of executive function ability | Baseline (at 7-10 months after start of therapy) and at 3 months after baseline
  To assess the impact of a computer-based working memory intervention, relative to standard of care, on additional performance- and rater-based measure of executive function. Executive function is measured as age-appropriate by the following: BRIEF-P (age 3 to <6 years), BRIEF (age 6 to <19 years) and BREIF-A (age ≥19 years). Connor's Parent Rating Scale, Third Edition (CPRS-III) will also be used for age 6 to <19 years, as well as CogState One-Back and Groton Maze tasks for age ≥5 years. T tests will be used to compare changes in executive function between the intervention and standard of care groups.
Change in measure of attention among 3 groups (working memory intervention + physical exercise intervention VS. working memory intervention alone VS. physical training intervention alone) | Baseline and at 3 months after baseline
  Working memory intervention baseline=7-10 months after on treatment. Physical exercise intervention baseline=at patient enrollment. Attention will be measured using different instruments as age appropriate: Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) for 3 to < 6 years (Digit Span Forward subtest), Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV) for 6 to < 17 years (Digit Span Forward subtest) or Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) for ≥17 years (Digit Span Forward subtest). We will also use Conners' Continuous Performance Test, Kiddie Version V.5 for 4 to < 6 years and Conner's Continuous Performance Test, Second Edition (CPT-II) for ≥6 years, in addition to Cog Stage for children ≥5 years (Detection and Identification tasks). ANOVA will be used to compare changes in memory among the groups. In addition, T-tests will be used to compare the combined intervention group to each of the other two groups.
Change in measure of processing speed among 3 groups (working memory intervention + physical exercise intervention VS. working memory intervention alone VS. physical training intervention alone) | Baseline and at 3 months after baseline
  Working memory intervention baseline=7-10 months after on treatment. Physical exercise intervention baseline=at patient enrollment. Cognitive processing speed function will be measured using the age-appropriate processing speed indices: WPPSI-IV which has two subsets: Bug Search and Cancellation, for 3 to < 6 years; WISC-IV which has two subsets: Coding and Symbol Search subtests, for 6 to < 17 years, and WAIS-IV which has two subsets: Coding and Symbol Search subtests, for ≥17 years. ANOVA will be used to compare changes in processing speed among the groups. In addition, T-tests will be used to compare the combined intervention group to each of the other two groups.
Change in measure of executive function among 3 groups (working memory intervention + physical exercise intervention VS. working memory intervention alone VS. physical training intervention alone) | Baseline and at 3 months after baseline
  Working memory intervention baseline=7-10 months after on treatment. Physical exercise intervention baseline=at patient enrollment. Executive function is measured as age-appropriate by the following: BRIEF-P (3 to <6 years), BRIEF (6 to <19 years) and BREIF-A (≥19 years). Connor's Parent Rating Scale, Third Edition (CPRS-III) will also be used for 6 to <19 years, as well as CogState One-Back and Groton Maze tasks for ≥5 years. ANOVA will be used to compare changes in executive function among the groups. In addition, T-tests will be used to compare the combined intervention group to each of the other two groups.
Change in measure of attention between participants who received computer-based intervention VS. those who did not | Baseline (at 7-10 months after on treatment) through 6 months after baseline.
  Attention will be measured using different instruments as age appropriate: Wechsler Preschool and Primary Scale of Intelligence, Fourth Edition (WPPSI-IV) for 3 to < 6 years (Digit Span Forward subtest), Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV) for 6 to < 17 years (Digit Span Forward subtest) or Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) for ≥17 years (Digit Span Forward subtest). We will also use Conners' Continuous Performance Test, Kiddie Version V.5 for 4 to < 6 years and Conner's Continuous Performance Test, Second Edition (CPT-II) for ≥6 years, in addition to Cog Stage for ≥5 years (Detection and Identification tasks). Differences between 6 months following assessment and immediate post-intervention testing, and difference between 6 months following assessment and pre-intervention testing, will be calculated for each subject and then group difference (intervention group vs. control group) will be examined using t-tests.
Change in measure of working memory between participants who received computer-based intervention VS. those who did not | Baseline (at 7-10 months after on treatment) through 6 months after baseline.
  To evaluate the maintenance of improvements in working memory three months following participation in the computer-based working memory intervention program. Memory will be measured using different instruments as age appropriate: CogStage for ≥5 years (Continuous Paired Associate Learning task), California Verbal Learning Test, Children's Version (CVLT-C) for 6 to < 17 years or California Verbal Learning Test, Second Edition (CVLT-II) for ≥17 years. The differences between six months following assessment and immediate post-intervention testing, as well as the difference between six months following assessment and pre-intervention testing, will be calculated for each subject and then the group difference (intervention group vs. control group) will be examined using t-tests.
Change in measure of processing speed between participants who received computer-based intervention VS. those who did not | Baseline (at 7-10 months after on treatment) through 6 months after baseline.
  To evaluate the maintenance of improvements on processing speed three months following participation in the computer-based working memory intervention program. Cognitive processing speed function will be measured using the age-appropriate processing speed indices: WPPSI-IV which has two subsets: Bug Search and Cancellation, for 3 to < 6 years; WISC-IV which has two subsets: Coding and Symbol Search subtests, for 6 to < 17 years, and WAIS-IV which has two subsets: Coding and Symbol Search subtests, for ≥17 years. The differences between six months following assessment and immediate post-intervention testing, as well as the difference between six months following assessment and pre-intervention testing, will be calculated for each subject and then the group difference (intervention group vs. control group) will be examined using t-tests.
Change in measure of executive function between participants who received computer-based intervention VS. those who did not | Baseline (at 7-10 months after on treatment) through 6 months after baseline.
  To evaluate the maintenance of improvements in executive function three months following participation in the computer-based working memory intervention program. Executive function is measured as age-appropriate by the following: BRIEF-P (3 to <6 years), BRIEF (6 to <19 years) and BREIF-A (≥19 years). Connor's Parent Rating Scale, Third Edition (CPRS-III) will also be used for 6 to <19 years, as well as CogState One-Back and Groton Maze tasks for ≥5 years. The differences between six months following assessment and immediate post-intervention testing, as well as the difference between six months following assessment and pre-intervention testing, will be calculated for each subject and then the group difference (intervention group vs. control group) will be examined using t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Gajjar, MD, Principal Investigator — St. Jude Children's Research Hospital; Giles Robinson, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (23):
- United States (14):
  - Lucille Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - Yale University, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Duke Children's Hospital and Health Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Cancer Center, Houston, Texas
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Melbourne, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- Starship Children's Hospital, Auckland, New Zealand

REFERENCES:
- [Derived] Khan RB, Patay Z, Klimo P, Huang J, Kumar R, Boop FA, Raches D, Conklin HM, Sharma R, Simmons A, Sadighi ZS, Onar-Thomas A, Gajjar A, Robinson GW. Clinical features, neurologic recovery, and risk factors of postoperative posterior fossa syndrome and delayed recovery: a prospective study. Neuro Oncol. 2021 Sep 1;23(9):1586-1596. doi: 10.1093/neuonc/noab030. PMID 33823018
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols